CLINICAL TRIAL: NCT07363395
Title: A Phase 1, First-in-human, Randomized, Double-blind, Placebo-controlled, Single and Multiple Ascending Dose Study to Assess the Safety, Tolerability, and Pharmacokinetics of ASCT-83 Subcutaneous Injection in Healthy Adults
Brief Title: Safety, Tolerability, and Pharmacokinetics of ASCT-83 in Healthy Adults
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Alcamena Stem Cell Therapeutics (Industry)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH); Congressionally Directed Medical Research Programs (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Treatment
Other Study IDs: ASCT-83-101; 1R44NS145934-01 (NIH); CDMRP-HT94252510912 (Other Grant/Funding Number: U.S. Army Medical Research Acquisition Activity (USAMRAA))
Record Dates: First submitted 2026-01-09; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2026-01

CONDITIONS: Neuropathic Pain
Keywords: Neuropathic Pain; Nerve Regeneration; Analgesic; CTDSP1 Inhibitor; REST (RE1-silencing transcription factor); Macrocyclic Peptide; Target Engagement; First-in-Human (FIH); SAD/MAD; Healthy Volunteers; Pharmacokinetics (PK); Diabetic Peripheral Neuropathy (DPN); Peripheral Nerve Injury (PNI)
MeSH Terms: conditions — Neuralgia; Peripheral Nerve Injuries

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (11):
- SAD-Placebo (Placebo Comparator): One dose of placebo solution administered as two subcutaneous injections of 1.5 ml (second injection within 10 minutes of the first)
  Interventions: Drug: Placebo
- SAD, ASCT-83 dose 1 (Experimental): Total dose: 0.5 mg ASCT-83. Administration: two 1.5 mL subcutaneous injections of 0.17 mg/mL (second injection within 10 minutes of the first)
  Interventions: Drug: ASCT-83
- SAD, ASCT-83 dose 2 (Experimental): Total dose: 1 mg ASCT-83. Administration: two 1.5 mL subcutaneous injections of 0.33 mg/mL (second injection within 10 minutes of the first)
  Interventions: Drug: ASCT-83
- SAD-ASCT dose 3 (Experimental): Total dose: 2 mg ASCT-83. Administration: two 1.5 mL subcutaneous injections of 0.67 mg/mL (second injection within 10 minutes of the first)
  Interventions: Drug: ASCT-83
- SAD-ASCT dose 4 (Experimental): Total dose: 4 mg ASCT-83. Administration: two 1.5 mL subcutaneous injections of 1.33 mg/mL (second injection within 10 minutes of the first)
  Interventions: Drug: ASCT-83
- SAD, ASCT-83 dose 5 (Experimental): Total dose: 7.5 mg ASCT-83. Administration: two 1.5 mL subcutaneous injections of 2.5 mg/mL (second injection within 10 minutes of the first)
  Interventions: Drug: ASCT-83
- SAD, ASCT-83 dose 6 (Experimental): Total dose: 10 mg ASCT-83. Administration: two 1.5 mL subcutaneous injections of 3.33 mg/mL (second injection within 10 minutes of the first)
  Interventions: Drug: ASCT-83
- MAD-Placebo (Placebo Comparator): Two daily subcutaneous injections of 1.5 ml placebo for 7 days, with the two daily injections given max 10 minutes apart.
  Interventions: Drug: Placebo
- MAD, ASCT-83 dose 1 (Experimental): Two daily subcutaneous injections of 1.5 ml of ASCT-83 for 7 days, with the two daily injections given max 10 minutes apart. Dose to be determined.
  Interventions: Drug: ASCT-83
- MAD, ASCT-83 dose 2 (Experimental): Two daily subcutaneous injections of 1.5 ml of ASCT-83 for 7 days, with the two daily injections given max 10 minutes apart. Dose to be determined.
  Interventions: Drug: ASCT-83
- MAD, ASCT-83 dose 3 (Experimental): Two daily subcutaneous injections of 1.5 ml of ASCT-83 for 7 days, with the two daily injections given max 10 minutes apart. Dose to be determined.
  Interventions: Drug: ASCT-83

INTERVENTIONS:
Drug: ASCT-83 — ASCT-83 is a 23-amino acid, macrocyclic peptide with a molecular weight of approximately 3 kilodaltons under development for the treatment of neuropathic pain (NeP).
  ASCT-83 25 mg/mL sterile solution for injection consists of 25 mg of ASCT-83 drug substance dissolved in 1 mL of histidine buffer. The product also contains mannitol to adjust the osmolarity of the final product. The product is stored at -20°C prior to dilution to achieve the target dose.
  Arms: MAD, ASCT-83 dose 1; MAD, ASCT-83 dose 2; MAD, ASCT-83 dose 3; SAD, ASCT-83 dose 1; SAD, ASCT-83 dose 2; SAD, ASCT-83 dose 5; SAD, ASCT-83 dose 6; SAD-ASCT dose 3; SAD-ASCT dose 4
Drug: Placebo — Placebo solution contaninig the same histidine buffer and mannitol concentrations as ASCT-83, with polyoxyl 35 castor oil (0.1% w/v) added to match the appearance of the active solution.
  Arms: MAD-Placebo; SAD-Placebo

SUMMARY:
The goal of this clinical trial is to learn if ASCT-83 is safe and well-tolerated and measure how ASCT-83 is absorbed, distributed, and eliminated from the body over time. The study will be conducted in healthy adults.

The main questions this study will answer are:

* Is ASCT-83 safe at clinical doses?
* Does ASCT-83 have side effects at clinical doses?
* How is ASCT-83 absorbed, distributed, and eliminated from the body? Researchers will compare ASCT-83 to a placebo (a look-alike substance that contains no drug).

The study has two parts: participants in Part 1 will receive only one dose of ASCT-83 or placebo participants in Part 2 will receive one dose of ASCT-83 or placebo a day for 7 days. Participants will visit the clinic to take ASCT-83 or placebo, to receive health checkups and undergo health tests. Participants in Part 1 will spend 5 days/4 nights in the clinic, participants in Part 2 will spend 11 days/10 nights in the clinic. In addition, there will be up to 3 outpatient visits.

The results of this study will help determine safe dose levels and support the design of future clinical trials.

DETAILED DESCRIPTION:
Seventy-two healthy participants will be randomized to the following groups:

* Part 1, Single Ascending Dose (SAD): Healthy adult participants (age 18-64, inclusive) will be enrolled in 6 dose cohorts: 0.5 mg, 1 mg, 2 mg, 4 mg, 7.5 mg, or 10 mg. Each cohort consists of 8 participants (6 ASCT-83, 2 placebo), totaling 48 participants.
* Part 2, Multiple Ascending Dose (MAD): 3 dose cohorts of 8 participants each (6 ASCT-83, 2 placebo), totaling 24 participants. Dosing and regimens for Part 2 will be determined following review of SAD data by the Data Safety Monitoring Committee (DSMC).

All doses (ASCT-83 or placebo) will be administered as two subcutaneous (SC) injections (arm or thigh), with the second injection occurring within 10 minutes of the first.

The first two participants in every cohort - one administered ASCT-83 and one administered placebo - will be the sentinel participants. In every cohort, the two sentinel participants must be observed for 72 hours before the rest of the cohort is dosed.

The maximum dose escalation increment between any two cohorts will be two-fold. The maximum daily dose will not exceed the maximum tolerated dose established in the SAD study.

Additional cohorts may be recruited based on the emerging safety, tolerability, and PK data.

ELIGIBILITY:
Inclusion Criteria:

To participate in the study, you must:

* be medically healthy based on medical history, physical exam, labs, and ECG
* be 18-64 years (inclusive)
* at screening, have a body mass index (BMI) > 19 to < 35 kg/m²
* be willing and able to understand and voluntarily sign an informed consent
* Female participants of childbearing potential (women who can become pregnant) must:

  1. agree to follow the study contraceptive requirements from screening through 28 days after the final dose of study drug.
  2. agree to undergo pregnancy testing, including a negative pregnancy test at screening and at admission.
  3. agree not to donate ova (eggs) from screening through 28 days after the final dose of study drug.
* Male participants must:

  1. have a vasectomy greater than 6 months prior to screening or be willing to follow the contraceptive requirements from screening through 90 days after final study drug administration
  2. agree to be willing to abstain from sperm donation from screening through 90 days after final study drug administration

Exclusion Criteria:

You cannot participate in the study if you:

* are a study site staff, Alcamena employee or immediate family member, or have participated in another clinical trial within 30 days or 5 half-lives of a prior investigational product.
* have evidence of liver disease or abnormal liver tests (ALT/AST, Alk Phos, GGT, or bilirubin > ULN); positive hepatitis B or C serology (people with Gilbert syndrome may be included).
* have a history of kidney disease, protein in the urine or reduced kidney function based on screening blood tests.
* have a history of cancer with active disease, suspected relapse, treatment within 6 months, or ongoing therapy affecting immune, liver, or kidney function.
* have a history of heart disease, including abnormal heart rhythm, heart attack, long QT syndrome, or abnormal heart rhythm findings on screening ECG, or a family history of sudden unexplained death.
* are currently receiving medications that affect or suppress the immune system, including steroids given by any route.
* have a known autoimmune condition (such as lupus, rheumatoid arthritis, sarcoidosis, or vitiligo), even if it is not being treated.
* have a positive HIV test at screening or a history of immune deficiency.
* have abnormal blood tests suggesting ongoing inflammation
* have an active infection or is currently being treated for an infection.
* have a skin condition that could interfere with study skin assessments (such as psoriasis).
* are allergic or sensitive to the study drug or its ingredients.
* have a history of alcohol or drug abuse or addiction within the past five years, have a positive drug or alcohol test at screening, or have smoked within one month before screening.
* have a serious mental health condition, such as major depression, schizophrenia, severe anxiety, eating disorders, severe attention deficit disorder, personality disorders, or suicidal thoughts or behavior within the past five years that could affect safety or study participation.
* have low blood pressure upon standing, defined as a significant drop in blood pressure when moving from lying down to standing during screening or baseline testing.
* have abnormally low white blood cell counts or neutrophil counts, unless this finding is due to a known benign condition such as benign ethnic neutropenia.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2026-10 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Incidence, severity and dose relationships of Treatment-Emergent Adverse Events (TEAEs) and non-TEAEs, Adverse Events of Special Interest (AESIs), Serious Adverse Events (SAEs), premature treatment and study discontinuation due to Adverse Events (AEs) | Single dose part of the study: from enrollment to 30-32 days after the end of treatment. Multiple dose part of the study: from enrollment to 36-38 days after the end of treatment.
  The investigator will assess and record information pertaining to the AE, which includes but is not limited to the following: date of onset, event diagnosis (when known) and/or signs and symptoms, duration, severity, seriousness (i.e. serious adverse event or not serious), expected/unexpected, and relationship to the study therapy or procedure, action(s) taken, and outcome. Severity grading: 1 Mild; asymptomatic or mild symptoms; clinical or diagnostic observations only; intervention not indicated.
  2 Moderate; minimal, local, or noninvasive intervention indicated; limiting age-appropriate instrumental ADL.
  3 Severe or medically significant but not immediately life-threatening; hospitalization or prolongation of hospitalization indicated; disabling; limiting self-care ADL.
  4 Life-threatening consequences; urgent intervention indicated. 5 Death related to AE.
Incidence and severity of changes in clinical safety parameters, including vital signs (including body weight), laboratory (including markers of inflammation), ECG results, and skin assessments (including injection site reactions). | Single dose part of the study: from enrollment to 30-32 days after the end of treatment. Multiple dose part of the study: from enrollment to 36-38 days after the end of treatment.
Incidence of suicidality | Single dose part of the study: from enrollment to 30-32 days after the end of treatment. Multiple dose part of the study: from enrollment to 36-38 days after the end of treatment.
  Suicide risk will be assessed through a questionnaire (Columbia-Suicide Severity Rating Scale (C-SSRS)). A score ≥4 is considered suicidal ideation.
Incidence and type of abnormal skin assessments, including injection-site reactions. | Single dose part of the study: from enrollment to 30-32 days after the end of treatment. Multiple dose part of the study: from enrollment to 36-38 days after the end of treatment.
  The FDA Toxicity Grading Scale (TGS) for injection/vaccine sites will be used: Mild/Grade 1, Moderate/Grade 2, Severe/Grade 3, Life-threatening/Grade 4.

SECONDARY OUTCOMES:
Area under the concentration-time curve from time zero to infinity (AUC0-inf) of ASCT-83 | SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose. MAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1; pre-dose on Days 3 to 7; 24, 36, 48, and 72 hours after the final dose on Day 7
  Plasma concentration of ASCT-83 will be measured following a single dose of ASCT-83 (SAD part of the study) or multiple doses of ASCT-83 (MAD part of the study) to characterize the total exposure to ASCT-83.
Area under the concentration-time curve from time zero to 24 h (AUC0-24h) of ASCT-83 | SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose. MAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1; pre-dose on Days 3 to 7; 24, 36, 48, and 72 hours after the final dose on Day 7
  Plasma concentration of ASCT-83 will be measured following a single dose of ASCT-83 (SAD part of the study) or multiple doses of ASCT-83 (MAD part of the study) to characterize exposure to ASCT-83 over the last 24 h dosing interval.
Peak plasma concentration (Cmax) of ASCT-83 | SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose. MAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1; pre-dose on Days 3 to 7; 24, 36, 48, and 72 hours after the final dose on Day 7
  Plasma concentration of ASCT-83 will be measured to characterize the peak concentration of ASCT-83 in the blood following either a single dose (SAD part of the study) or multiple doses (MAD part of the study) of ASCT-83.
Time to reach maximum plasma concentration (Tmax) of ASCT-83 | SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose. MAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1; pre-dose on Days 3 to 7; 24, 36, 48, and 72 hours after the final dose on Day 7
  Plasma concentrations of ASCT-83 will be measured to determine the time at which the highest concentration of ASCT-83 is reached after either a single dose (SAD part of the study) or multiple doses of ASCT-83 (MAD part of the study).
Terminal elimination half-life (t½) of ASCT-83 | SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose. MAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1; pre-dose on Days 3 to 7; 24, 36, 48, and 72 hours after the final dose on Day 7
  Concentrations of ASCT-83 in plasma will be measured to determine the time required for the drug concentration to decrease to half of its initial amount. Plasma concentrations will be measured both in the single dose (SAD) and the multiple dose (MAD) part of the study.
Apparent clearance (CL/F) of ASCT-83 | SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose. MAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1; pre-dose on Days 3 to 7; 24, 36, 48, and 72 hours after the final dose on Day 7
  Plasma clearance of ASCT-83 will be measured after both a single dose (SAD part of the study) and multiple doses (MAD part of the study) of ASCT-83.
Apparent volume of distribution (Vz/F) of ASCT-83 | SAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24, 36, 48, 72 hours post-dose. MAD: pre-dose, 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 10, 12, 24 hours post-dose on Day 1; pre-dose on Days 3 to 7; 24, 36, 48, and 72 hours after the final dose on Day 7
  The distribution of ASCT-83 in the body (whether it stays in the blood or it spreads to the rest of the body) will be measured after a single dose (SAD part of the study) or multiple doses (MAD part of the study) of ASCT-83.
Amount of ASCT-83 excreted in urine | Pre-dose, then at 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours, 24-36 hours, 36-48 hours, 48-60 hours, 60-72 hours post-dose.
  Amount of ASCT-83 excreted in urine will be measured after a single dose of ASCT-83 (SAD part of the study).
Fraction of ASCT-83 excreted in urine unchanged | Pre-dose, then at 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours, 24-36 hours, 36-48 hours, 48-60 hours, 60-72 hours post-dose.
  The proportion of ASCT-83 that is eliminated in urine in its original, active form will be measured after a single dose of ASCT-83 (SAD part of the study).
Renal clearance (CLR) of ASCT-83 | Pre-dose, then at 0-4 hours, 4-8 hours, 8-12 hours, 12-24 hours, 24-36 hours, 36-48 hours, 48-60 hours, 60-72 hours post-dose.
  The amount of ASCT-83 excreted in the urine during an interval of time will be measured after a single dose of ASCT-83 (SAD part of the study).
Incidence of anti-drug antibodies (ADA) and titers (in ADA positive participants). | Prior to initiation of dosing on Day 1, and on Days 7, 14, 25, 37.

OTHER OUTCOMES:
Quantification of Pharmacodynamic (PD) Biomarkers of Target Engagement: SMAD1/5/8 | SAD: pre-dose on Day 1 and 24 hours after dosing (Day 2). MAD: pre-dose on Day 1 and 4 hours after the third and last dosing.
  Single dose part of the study (SAD): Phospho-SMAD1/5/8 levels will be measured in Peripheral Blood Mononuclear Cells (PBMCs) following ex vivo BMP4 stimulation. Multiple dose part of the study (MAD): total SMAD1/5/8 depletion will be measured in unstimulated PBMC lysates.
Quantification of Pharmacodynamic (PD) Biomarkers of Target Engagement: BDNF | SAD: pre-dose on Day 1 and 24 hours after dosing (Day 2). MAD: pre-dose on Day 1 and 4 hours after the third and last dosing.
  The change from baseline levels in the amount of Brain-Derived Neurotrophic Factor (BDNF) circulating in the blood will be measured in plasma after a single dose of ASCT-83.

CONTACTS AND LOCATIONS:
Overall Officials: Edmund Nesti, PhD, Study Director — Alcamena Stem Cell Therapeutics; Trisha Shamp, PhD, PA-C, ECG-BA, CVPA-BC, Principal Investigator — Nucleus Network

IPD SHARING:
Plan to Share IPD: No
Participant data is restricted to the Sponsor and oversight bodies (FDA/DoD)